CLINICAL TRIAL: NCT03029702
Title: Metabolic Analysis for Treatment Choice in Gestational Diabetes Mellitus
Acronym: MATCh-GDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maisa N. Feghali, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Maisa N. Feghali, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO16100499; K23HD092893 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes; Diabetes, Gestational; Pregnancy in Diabetes
Keywords: Gestational diabetes; Diabetes in pregnancy; Insulin resistance; Insulin secretion deficiency
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics; Insulin Resistance | interventions — Insulin; Glyburide; Metformin

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Study team members assessing delivery outcomes will be masked to the participant's study assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Participants will undergo standard counseling and be prescribed a treatment for their GDM. Treatments include insulin, glyburide, and metformin.
  Interventions: Drug: Insulin; Drug: Glyburide; Drug: Metformin
- Individualized Treatment (Active Comparator): Participants will undergo standard counseling and be matched to therapy based on their GDM mechanism. Treatments include insulin, glyburide, and metformin.
  Interventions: Drug: Insulin; Drug: Glyburide; Drug: Metformin

INTERVENTIONS:
Drug: Insulin — Insulin will be used for GDM treatment
Drug: Glyburide — Glyburide will be used for GDM treatment
Drug: Metformin — Metformin will be used for GDM treatment

SUMMARY:
Gestational diabetes (GDM) is a significant clinical and public health burden, affecting over 400,000 pregnant women in the United States each year. Without adequate treatment, women with GDM and their infants are at risk for substantial morbidity. Because of this, experts recommend treatment focused on normalization of hyperglycemia to improve outcomes. However, providers have limited capacity to predict which treatment will achieve glycemic goals. This results in a choice based on provider and patient preference and a trial and error approach, which can create delays in glycemic control within the short (8-10 weeks) window between diagnosis and delivery. Maternal and fetal morbidity may be related to a mismatch between glycemic pathophysiology and the mechanism of action of glucose-lowering agents. In fact, GDM is heterogeneous, with predominant insulin resistance (IR) in 50%, insulin secretion deficit (ISD) in 30%, and a combination of both in 20% of women as underlying mechanisms of hyperglycemia. This variation in GDM pathophysiology and clinical outcomes supports the use of an individualized treatment approach. The overall goal of this project is to investigate an individualized treatment approach for GDM where treatment is based on each woman's GDM mechanism. The study will employ the same treatment in both arms, but choice of treatment will differ based on study arm (matched or unmatched to GDM mechanism).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women beyond 24 weeks of gestation who are scheduled for a 3-hour oral glucose tolerance test.

Exclusion Criteria:

* Fetal anomaly
* Pregestational diabetes
* GDM diagnosis without a 3-hour OGTT
* Multifetal gestation
* Treatment with non-inhaled steroids within 7 days
* Allergy to glyburide, metformin or sulfa
* History of severe pulmonary (pulmonary requirement for oxygen therapy or daily treatment for restrictive of obstructive pulmonary disease)
* Hepatic (LFT's greater than two times of upper normal range)
* Renal (serum creatinine higher than 1.2 mg/dL) disease
* History of heart failure or myocardial infarction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maisa N Feghali, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Individualized Treatment
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Individualized Treatment | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.90 (5.9) | 30.91 (6.6) | 30.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 14 | 13 | 27
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Who Are Eligible, Screened, Enroll and Remain in the Study
Description: Proportion of women who are eligible, screened, enrolled and remain in the study
Time Frame: Through study completion, an average of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 25 | 26
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.9, Fisher Exact

2. Primary Outcome: Proportion of Participants Who Report Suitability of the Study Procedures
Description: Suitability of the study procedures and interventions to participants assessed through one-on-one qualitative interview
Time Frame: Through study completion, an average of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 24 | 25
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.8, Fisher Exact

3. Secondary Outcome: Proportion of Participants With Consistent GDM Mechanism Before and and After Treatment Initiation
Time Frame: 2 weeks after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 22 | 21
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.9, Fisher Exact

4. Secondary Outcome: Proportion of Women Who Remain on Same Treatment During Study
Time Frame: Through study completion, an average of 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 25 | 26
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.9, Fisher Exact

5. Secondary Outcome: Maternal Glucose Control
Description: >50% fasting below 95 and 1 hour postprandial < 140 during the 4 weeks before delivery
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 20 | 22
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.8, Fisher Exact

6. Secondary Outcome: Proportion of Participants Who Deliver by Primary Cesarean
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 9 | 11
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.6, Chi-squared

7. Secondary Outcome: Proportion of Participants Who Developed Hypertensive Diseases in Pregnancy
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
Participants | 4 | 3
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.8, Chi-squared

8. Secondary Outcome: Birthweight
Time Frame: Delivery
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 27 | 27
g | 332.5 (376.7) | 3445.4 (627.2)
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p = 0.7, t-test, 2 sided

9. Secondary Outcome: Neonatal Lean Body Mass
Time Frame: Within 72 hours of delivery
Population: Unable to collect neonatal data due to lack of staffing availability
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Cord Blood Glucose
Time Frame: Delivery
Population: Samples unavailable for analysis due to freezer storage malfunction
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Cord Blood C-peptide
Time Frame: Delivery
Population: Samples unavailable for analysis due to freezer storage malfunction
Arm/Group | Usual Care | Individualized Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study participation ~ 6 months
Arm/Group | Usual Care | Individualized Treatment
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03029702/Prot_SAP_002.pdf